CLINICAL TRIAL: NCT02084615
Title: A Prospective, Nonrandomized, Study Comparing the Use of Aspirin and Intraoperative Blood Loss and Postoperative Complications Following Open Inguinal Hernia Repair.
Brief Title: Prospective Study Investigating Aspirin and Intraoperative Blood Loss and Complications Following Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jesse Brown VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joseph Vitello, MD, Interim Chief of Surgical Services, Jesse Brown VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0976
Record Dates: First submitted 2014-03-09; First posted 2014-03-12 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Hernia, Inguinal; Postoperative Complications; Postoperative Hemorrhage
Keywords: Aspirin; Postoperative hemorrhage; Inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal; Postoperative Complications; Postoperative Hemorrhage | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 81mg aspirin (Experimental): This arm will include perioperative 81 mg of aspirin.
  Interventions: Drug: Aspirin
- 325mg aspirin (Experimental): Subjects will be taking 325mg of aspirin.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Subjects will undergo open inguinal hernia repairs while taking their normal dose of 81mg, 325mg, or no aspirin
  Other Names: acetylsalicylic acid

SUMMARY:
The purpose of this study is to determine whether aspirin taken in the perioperative period will increase the blood loss associated with open inguinal hernia repairs. A secondary purpose of this study is to determine if the aspirin administered in the perioperative period increases the risk of complications associated with open inguinal hernia repairs.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, study which compares the use of 81mg of aspirin, 325mg of aspirin or no aspirin in adult men undergoing an open tension free mesh inguinal hernia repair. Subjects currently taking 81mg or 325mg of aspirin will undergo inguinal hernia repair without having their medications stopped. Patient not currently taking aspirin will act as controls. Intraoperative blood loss will be measured utilizing a gravimetric method by weighing surgical sponges before and after use. Subjects will be followed for thirty days postoperatively and be evaluated for bleeding complications. The specific complications include wound or scrotal hematomas, return to the operating room within 72 hour for bleeding, wound infection, early recurrent hernia, excessive wound ecchymosis.

ELIGIBILITY:
Inclusion Criteria:

* adult male veterans ages 18-99
* inguinal hernia
* subjects currently taking 81mg, 325mg or no aspirin

Exclusion Criteria:

* recurrent hernia
* "giant" hernia
* women
* International Normalized Ratio > 1.7
* Hemophilia or other know congenital bleeding disorder
* Cirrhosis of hepatitis with coagulopathy
* Thrombocytopenia with platelet counts < 100,000
* Subjects currently on Coumadin or other platelet inhibitors

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | intraoperative only
  intraoperative blood loss will be accurately measured among the three arms of the study

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 30 days post operative
  Subjects will be followed for 30 days post-operatively for bleeding complications such as early return to the operating room to control bleeding, wound hematoma, scrotal hematoma, wound infection, early hernia recurrence, or excessive wound ecchymosis

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Vitello, MD, Principal Investigator — Jesse Brown VA Medical Center
Locations (1):
- Jesse Brown VA Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Antolovic D, Rakow A, Contin P, Ulrich A, Rahbari NN, Buchler MW, Weitz J, Koch M. A randomised controlled pilot trial to evaluate and optimize the use of anti-platelet agents in the perioperative management in patients undergoing general and abdominal surgery--the APAP trial (ISRCTN45810007). Langenbecks Arch Surg. 2012 Feb;397(2):297-306. doi: 10.1007/s00423-011-0867-7. Epub 2011 Nov 3. PMID 22048442
- [Background] Binhas M, Salomon L, Roudot-Thoraval F, Armand C, Plaud B, Marty J. Radical prostatectomy with robot-assisted radical prostatectomy and laparoscopic radical prostatectomy under low-dose aspirin does not significantly increase blood loss. Urology. 2012 Mar;79(3):591-5. doi: 10.1016/j.urology.2011.11.031. PMID 22386405
- [Background] Burger W, Chemnitius JM, Kneissl GD, Rucker G. Low-dose aspirin for secondary cardiovascular prevention - cardiovascular risks after its perioperative withdrawal versus bleeding risks with its continuation - review and meta-analysis. J Intern Med. 2005 May;257(5):399-414. doi: 10.1111/j.1365-2796.2005.01477.x. PMID 15836656
- [Background] Chechik O, Goldstein Y, Behrbalk E, Kaufman E, Rabinovich Y. Blood loss and complications following carotid endarterectomy in patients treated with clopidogrel. Vascular. 2012 Aug;20(4):193-7. doi: 10.1258/vasc.2011.oa0336. Epub 2012 May 10. PMID 22577162
- [Background] Gerstein NS, Schulman PM, Gerstein WH, Petersen TR, Tawil I. Should more patients continue aspirin therapy perioperatively?: clinical impact of aspirin withdrawal syndrome. Ann Surg. 2012 May;255(5):811-9. doi: 10.1097/SLA.0b013e318250504e. PMID 22470078
- [Background] Kang SB, Cho KJ, Moon KH, Jung JH, Jung SJ. Does low-dose aspirin increase blood loss after spinal fusion surgery? Spine J. 2011 Apr;11(4):303-7. doi: 10.1016/j.spinee.2011.02.006. PMID 21474081
- [Background] Leyh-Bannurah SR, Hansen J, Isbarn H, Steuber T, Tennstedt P, Michl U, Schlomm T, Haese A, Heinzer H, Huland H, Graefen M, Budaus L. Open and robot-assisted radical retropubic prostatectomy in men receiving ongoing low-dose aspirin medication: revisiting an old paradigm? BJU Int. 2014 Sep;114(3):396-403. doi: 10.1111/bju.12504. Epub 2014 Jul 15. PMID 24127902
- [Background] Madan GA, Madan SG, Madan G, Madan AD. Minor oral surgery without stopping daily low-dose aspirin therapy: a study of 51 patients. J Oral Maxillofac Surg. 2005 Sep;63(9):1262-5. doi: 10.1016/j.joms.2005.05.164. PMID 16122588
- [Background] Manning BJ, O'Brien N, Aravindan S, Cahill RA, McGreal G, Redmond HP. The effect of aspirin on blood loss and transfusion requirements in patients with femoral neck fractures. Injury. 2004 Feb;35(2):121-4. doi: 10.1016/s0020-1383(03)00073-1. PMID 14736467
- [Background] Ono K, Idani H, Hidaka H, Kusudo K, Koyama Y, Taguchi S. Effect of aspirin continuation on blood loss and postoperative morbidity in patients undergoing laparoscopic cholecystectomy or colorectal cancer resection. Surg Laparosc Endosc Percutan Tech. 2013 Feb;23(1):97-100. doi: 10.1097/SLE.0b013e318278cdf8. PMID 23386161
- [Background] Oscarsson A, Gupta A, Fredrikson M, Jarhult J, Nystrom M, Pettersson E, Darvish B, Krook H, Swahn E, Eintrei C. To continue or discontinue aspirin in the perioperative period: a randomized, controlled clinical trial. Br J Anaesth. 2010 Mar;104(3):305-12. doi: 10.1093/bja/aeq003. PMID 20150346
- [Background] Partridge CG, Campbell JH, Alvarado F. The effect of platelet-altering medications on bleeding from minor oral surgery procedures. J Oral Maxillofac Surg. 2008 Jan;66(1):93-7. doi: 10.1016/j.joms.2005.11.055. PMID 18083421
- [Background] Zigdon H, Levin L, Filatov M, Oettinger-Barak O, Machtei EE. Intraoperative bleeding during open flap debridement and regenerative periodontal surgery. J Periodontol. 2012 Jan;83(1):55-60. doi: 10.1902/jop.2011.110182. Epub 2011 May 12. PMID 21563946